CLINICAL TRIAL: NCT02063399
Title: Prospective 20,000-person Nasopharyngeal Carcinoma (NPC) Screening Programme Using Plasma Epstein-Barr Virus (EBV) DNA Analysis
Brief Title: Prospective Nasopharyngeal Carcinoma Screening Using Plasma Epstein-Barr Virus DNA Analysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Allen Chan, Professor, Chinese University of Hong Kong
Other Study IDs: CU-ChemPath-001
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: NPC; Cancer screening; Plasma EBV DNA
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples are retended for future study to evaluate the accuracy of sequencing-based biomarkers
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if the screening of nasopharyngeal carcinoma using plasma Epstein-Barr virus DNA analysis would result in the detecting NPC cases at earlier stages and improve survival.

DETAILED DESCRIPTION:
Epstein-Barr virus (EBV) infection is an important etiological factor for nasopharyngeal carcinoma (NPC). In a pilot study, we have shown that the analysis of Epstein-Barr virus (EBV) DNA in blood can detect early and asymptomatic NPC. However, it is unlcear if NPC screening can improve the prognosis of the screened NPC subjects.

20,000 male subjects aged from 40 to 62 will be recruited because the incidence of NPC is higher in this target group. Twenty millilitres of venous blood will be collected from each subject at enrolment for plasma EBV DNA analysis.

Subjects who have initial positive results for plasma EBV DNA will have another testing at approximately 4 weeks. Subjects who have persistently positive results for the two plasma EBV DNA analyses will be investigated using nasal endoscopic examination and MRI of the nasopharynx.

After the initial screening, all participants will be phone interviewed yearly to update their cancer status.

A second round of screening will be carried out at 3 to 5 years after the initial round of screening. Subjects will be screened with plasma EBV DNA as in the first round of screening. Subjects with initial positive results will be retested and those with persistently positive results will be investigated using nasal endoscopic examination and MRI of the nasopharynx.

ELIGIBILITY:
Inclusion Criteria:

* age 40 to 62 years
* ethnic Chinese
* male

Exclusion Criteria:

* history of nasopharyngeal carcinoma
* currently having a malignant disease
* active autoimmune disease
* HIV infection
* on systemic steroid treatment
* on immunosuppressant treatment

Ages: 40 Years to 62 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male Hong Kong residents of Chinese ethnicity
Sampling Method: Non-Probability Sample
Enrollment: 20302 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Stage distribution of nasopharyngeal carcinoma at the time of diagnosis | 3 years
  All the participants will be subjected to the screening of nasopharyngeal carcinoma (NPC) at the time of recruitment using plasma EBV DNA analysis. Subjects with positive results will be investigated using endoscopic examination and MRI. If the subject is confirmed of having NPC, the stage of the disease would be recorded.

SECONDARY OUTCOMES:
Incidence of nasopharyngeal carcinoma in screened negative group | 5 years
  Participants who are screened negative will be followed up yearly for 5 years after the screening. The incidence of NPC will be recorded.
Relative risk of developing nasopharyngeal carcinoma for subjects with positive test results | 5 years
  The relative risk of developing nasopharyngeal carcinoma for subjects with negative, transiently positive and persistently positive plasma Epstein-Barr virus DNA at enrolment will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-chee Allen Chan, MD, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chan KC, Hung EC, Woo JK, Chan PK, Leung SF, Lai FP, Cheng AS, Yeung SW, Chan YW, Tsui TK, Kwok JS, King AD, Chan AT, van Hasselt AC, Lo YM. Early detection of nasopharyngeal carcinoma by plasma Epstein-Barr virus DNA analysis in a surveillance program. Cancer. 2013 May 15;119(10):1838-44. doi: 10.1002/cncr.28001. Epub 2013 Feb 21. PMID 23436393
- [Background] Lo YM, Chan LY, Lo KW, Leung SF, Zhang J, Chan AT, Lee JC, Hjelm NM, Johnson PJ, Huang DP. Quantitative analysis of cell-free Epstein-Barr virus DNA in plasma of patients with nasopharyngeal carcinoma. Cancer Res. 1999 Mar 15;59(6):1188-91. PMID 10096545
- [Derived] Chan KCA, Lam WKJ, King A, Lin VS, Lee PPH, Zee BCY, Chan SL, Tse IOL, Tsang AFC, Li MZJ, Jiang P, Ai QYH, Poon DMC, Au KH, Hui EP, Ma BBY, Van Hasselt AC, Chan ATC, Woo JKS, Lo YMD. Plasma Epstein-Barr Virus DNA and Risk of Future Nasopharyngeal Cancer. NEJM Evid. 2023 Jul;2(7):EVIDoa2200309. doi: 10.1056/EVIDoa2200309. Epub 2023 Jun 27. PMID 38320164
- [Derived] Chan KCA, Woo JKS, King A, Zee BCY, Lam WKJ, Chan SL, Chu SWI, Mak C, Tse IOL, Leung SYM, Chan G, Hui EP, Ma BBY, Chiu RWK, Leung SF, van Hasselt AC, Chan ATC, Lo YMD. Analysis of Plasma Epstein-Barr Virus DNA to Screen for Nasopharyngeal Cancer. N Engl J Med. 2017 Aug 10;377(6):513-522. doi: 10.1056/NEJMoa1701717. PMID 28792880